CLINICAL TRIAL: NCT03613727
Title: Therapeutic Use of Intravenous Vitamin C in Allogeneic Stem Cell Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17-13299; NCI-2018-01502 (Other: NCI CTRP)
Record Dates: First submitted 2018-07-27; First posted 2018-08-03 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Lymphoid Leukemia; Myeloid Leukemia; Monocytic Leukemia; Myelodysplasia
Keywords: Vitamin C; Hematopoietic cell transplant (HCT); Non-relapse mortality; Graft versus Host Disease (GVHD)
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Myeloid; Leukemia, Monocytic, Acute; Anemia, Refractory, with Excess of Blasts; Graft vs Host Disease | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IV Vitamin C followed by oral Vitamin C (Experimental): All study participants will receive the same treatment. Each participant will be given intravenous, which means by vein (IV), vitamin C three times a day for 14 days. Then participants will take vitamin C orally (by mouth in pill form) twice a day each day until 6 months after transplant. The treatment is IV vitamin C 50 mg/kg/day. After completion of the IV vitamin C doses, oral vitamin C 500 mg twice each day.
  Interventions: Drug: Intravenous (IV) and oral Vitamin C

INTERVENTIONS:
Drug: Intravenous (IV) and oral Vitamin C — Intravenous (IV) vitamin C 50 mg/kg/day divided in 3 doses beginning on posttransplant Day +1 and continuing through Day +14; each dose (16.7 mg/kg) given in 50 mL of 5% dextrose and water over 30 minutes every 8 hours
  • After completion of the IV vitamin C doses, oral vitamin C 500 mg twice each day beginning on Day +15 and continuing until Day +180
  Other Names: L-ascorbic acid

SUMMARY:
This phase 2 trial studies the effect of intravenous (IV) vitamin C repletion after myeloablative allogeneic stem cell transplant.

DETAILED DESCRIPTION:
Vitamin C is a nutritional supplement that can help fight inflammation. Most patients who have a stem cell transplant have lower than normal levels of vitamin C in their blood. Patients will receive intravenous Vitamin C the day after transplant for two weeks, followed by oral vitamin C until six months after transplant. The effect of the Vitamin C on non-relapse mortality (NRM), time to engraftment, rate of acute graft-versus-host disease and to characterize the safety and tolerability of the vitamin C regimen.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet all of the following inclusion criteria to be eligible to participate in the study:

1. Any of the following hematological malignancies:

   * Acute lymphoblastic leukemia
   * Acute myelogenous leukemia
   * Chronic myelogenous leukemia
   * Myelodysplasia
2. Candidate for hematopoietic cell transplant (HCT) Note: Patients with or without previous myeloablative autologous transplant are eligible.
3. human leukocyte antigen (HLA) matched stem cell donor, either related (6/6 or 5/6 loci matched) or unrelated (8/8 or 7/8 loci matched)
4. Stem cell graft from either bone marrow or peripheral blood
5. Negative serology for HIV
6. Age ≥ 18 to < 78 years of age
7. Karnofsky Performance Status of 70-100%
8. Women who are not postmenopausal or have not undergone hysterectomy must have a documented negative serum pregnancy test per standard Massey Cancer Center- Virginia Commonwealth University Health System (MCC-VCUHS) Bone Marrow Transplant (BMT) Program guidelines
9. Ability to understand and the willingness to sign a written informed consent document. Note: The consent form must be signed and dated prior to initiation of stem cell transplant (SCT) preparative treatments.

Exclusion Criteria:

* A patient who meets any of the following exclusion criteria is ineligible to participate in the study.

  1. Known allergy to vitamin C
  2. Inability to swallow oral medication
  3. Known or suspected malabsorption condition or obstruction
  4. G6PDH deficiency
  5. Uncontrolled viral, fungal, or bacterial infection
  6. Active meningeal or central nervous system disease
  7. Alternative hematopoietic cell transplant (HCT) including haplo-identical and umbilical cord transplants
  8. Non-myeloablative conditioning defined as total body irradiation (TBI) < 2 centigray (cGy)
  9. Pregnancy or breastfeeding
  10. Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Clark, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/ Massey Cancer Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants were consented and enrolled, but were not eligible to start treatment
Groups:
- IV Vitamin C Followed by Oral Vitamin C: All study participants will receive the same treatment. Each participant will be given intravenous, which means by vein (IV), vitamin C three times a day for 14 days. Then participants will take vitamin C orally (by mouth in pill form) twice a day each day until 6 months after transplant. The treatment is IV vitamin C 50 mg/kg/day. After completion of the IV vitamin C doses, oral vitamin C 500 mg twice each day.
  Intravenous (IV) and oral Vitamin C: Intravenous (IV) vitamin C 50 mg/kg/day divided in 3 doses beginning on posttransplant Day +1 and continuing through Day +14; each dose (16.7 mg/kg) given in 50 mL of 5% dextrose and water over 30 minutes every 8 hours
  • After completion of the IV vitamin C doses, oral vitamin C 500 mg twice each day beginning on Day +15 and continuing until Day +180
Period: Overall Study
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Number analyzed (Participants) | 55
Age, Customized [Count of Participants; unit: Participants]
  18 - 21 years | 1
  22 - 29 years | 2
  30 - 39 years | 7
  40 - 49 years | 5
  50 - 59 years | 21
  60 - 69 years | 18
  70 - 79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 49
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients That Experience Non-relapse Mortality (NRM)
Description: To determine the effect of parenteral vitamin C on non-relapse mortality (NRM) at one year following myeloablative allogeneic HCT. Non-relapse mortality is defined as defined as mortality from complications of HCT but not tumor relapse, is usually from graft versus host disease (GVHD), infection, or organ failure.
Time Frame: 1 year following myeloablative allogeneic hematopoietic cell transplant (HCT)
Measure: Count of Participants; unit: Participants
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Number analyzed (Participants) | 55
Participants | 5

2. Secondary Outcome: Time From Transplant to Engraftment
Description: To determine the effect of the vitamin C regimen on the time to hematopoietic engraftment.
Time Frame: 30 Days after myeloablative allogeneic hematopoietic cell transplant (HCT)
Measure: Median (Full Range); unit: Number of Days to engraftment
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Number analyzed (Participants) | 55
Number of Days to engraftment | 12 [9 to 15]

3. Secondary Outcome: To Determine the Effectiveness of Reducing Acute Graft Versus Host Disease (aGVHD)
Description: Percentage of patients with a diagnosis of acute GVHD
Time Frame: 0 - 180 days after myeloablative allogeneic HCT
Measure: Number; unit: percentage of participants
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Number analyzed (Participants) | 55
percentage of participants | 33

4. Secondary Outcome: Determine Related to Vitamin C Therapy Adverse Events (AEs) Reported Using Criteria in the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0)
Description: The number of participants who have adverse events related to Vitamin C therapy
Time Frame: Within first 30 days of myeloablative allogeneic HCT
Population: No participants had adverse events related to Vitamin C therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
Number analyzed (Participants) | 55
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 0 through Day 180.
Description: Adverse Events (AEs) >/= grade 3 regardless of expectedness or attribution were recorded
Arm/Group | IV Vitamin C Followed by Oral Vitamin C
All-Cause Mortality (participants affected / at risk) | 23/55
Serious Adverse Events (participants affected / at risk) | 40/55
Other Adverse Events (participants affected / at risk) | 55/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Vitamin C Followed by Oral Vitamin C (N=55)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Optic Nerve Disorder (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Sinusoidal obstruction syndrome (Hepatobiliary disorders) | 2 (2)
Catheter Related Infection (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Viremia (Infections and infestations) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Suicidial Ideation (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3)
Creatinie Increased (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Vitamin C Followed by Oral Vitamin C (N=55)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4)
Heart Failure (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Optic Nerve Disorder (Eye disorders) | 1 (1)
Vision Decreased (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 14 (17)
Nausea (Gastrointestinal disorders) | 5 (5)
Mucositis Oral (Gastrointestinal disorders) | 20 (20)
Small Intestinal Mucositis (Gastrointestinal disorders) | 8 (8)
Fatigue (General disorders) | 1 (1)
fever (General disorders) | 1 (1)
Sinusoidal Obstruction Syndrome (Hepatobiliary disorders) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Epstein-Barr Virus Infection Reactivation (Infections and infestations) | 9 (9)
Cytomegalovirus Infection Reactivation (Infections and infestations) | 14 (14)
Enterocolitis Infection Reactivation (Infections and infestations) | 1 (1)
Fungemia (Infections and infestations) | 1 (1)
Herpes Simplex Reactivation (Infections and infestations) | 1 (1)
Lung Infection (Infections and infestations) | 5 (7)
Sepsis (Infections and infestations) | 11 (12)
Skin Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 7 (7)
Viremia (Infections and infestations) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Blood Bilirubin Increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (10)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Weakness Lower Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Seizure (Nervous system disorders) | 1 (1)
Spinal Cord Compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypotension (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 2 (2)
Suicidial Ideation (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03613727/Prot_SAP_001.pdf
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03613727/ICF_000.pdf